CLINICAL TRIAL: NCT05307731
Title: Fingolimod for Type 2 Diabetes Mellitus: a Pilot, Prospective, Randomized, and Open Label Single-center Study
Brief Title: Fingolimod for Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, chief, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y(2021)071
Record Dates: First submitted 2022-03-21; First posted 2022-04-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fingoland group (Experimental): The patients of this group were treated with Fingolimod 0.5mg per day, in addition to guideline based treatment.
  Interventions: Drug: Fingolimod; Drug: guideline-based treatment for DM
- Control group (Active Comparator): The patients of this group were treated with diabetes drugs based on guideline
  Interventions: Drug: guideline-based treatment for DM

INTERVENTIONS:
Drug: Fingolimod — 0.5mg daily for 90-180 days, in addition to guideline-based treatment for DM
  Arms: Fingoland group
Drug: guideline-based treatment for DM — guideline-based treatment for DM

SUMMARY:
The aim of this study is to explore the efficacy and safety of Fingoland in the treatment of type 2 diabetes. A total of 40 patients were randomly divided into two groups. One group was treated with fingolimod, another group was given guideline based treatment. The changes of islet function in patients with glycosylated hemoglobin, insulin and C-peptide were observed .

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old;
2. clinically diagnosed type 2 diabetes.
3. Glycosylated hemoglobin: 6.5% - 9.5%;
4. No drug treatment or only one oral hypoglycemic drug within 6 months;
5. Fasting blood glucose: < 13.9mmol/l for those without medication, or < 13.3mmol/l for those with medication;
6. if the antidiabetic drugs are taken, the dosage and the drug must be stable in the past 3 months.
7. Body mass index (BMI) ≤ 45 kg / m2;
8. Sign informed consent

Exclusion Criteria:

1. patients with type 1 diabetes;
2. diabetic complications (ketoacidosis, hypertonic state, lactic acidosis).
3. Allergic to the study drug;
4. Abnormal liver and kidney function (transaminase greater than 2.5 times the upper limit of normal value; creatinine greater than 133umol / L);
5. Complicated with other serious organ diseases;
6. Recent disease history (within the past 6 months): myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or class III / IV heart failure;
7. Presence or history of mobitz type II second or third degree AV block or sick sinus syndrome, unless the patient has a pacemaker;
8. Baseline QT interval extension (male > 450ms or female > 460ms);
9. Treatment with class IA or class III antiarrhythmic drugs;
10. Patients with systemic infection (including but not limited to bacteria, fungi, viruses, etc.);
11. Participating in other clinical trials within 3 months;
12. Other circumstances that the investigator considers unsuitable for participating in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
The changes of glycosylated hemoglobin, compared with baseline | 180 days

SECONDARY OUTCOMES:
The changes of glycosylated hemoglobin, compared with baseline | 90 days, 120 days
The changes of treatment drugs, compared with baseline | 90 days, 120 days, 180 days
  including drug numbers and doses
The changes of 2-hour postprandial blood glucose, compared with baseline | 30 days, 90 days, 120 days, 180 days
The changes of fasting blood glucose, compared with baseline | 30 days, 90 days, 120 days, 180 days
Beta cell function, compared with baseline | 30 days, 90 days, 120 days, 180 days
  an oral glucose tolerance tests(OGTT) will be used to assess beta cell function.
The changes of insulin, compared with baseline | 30 days, 90 days, 120 days, 180 days
The changes of C-peptide, compared with baseline | 30 days, 90 days, 120 days, 180 days
any adverse events | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: HuiSheng Chen, Ph.D, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China